CLINICAL TRIAL: NCT03349437
Title: Pilot Study to Assess the Effect of Providing Intermittent Positive Airway Pressure in COPD Patients in Order to Relieve Their Exertion Related Shortness of Breath
Brief Title: Vitabreath Pilot in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRC-17007-VBIDEPILOT-PN
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2019-04-16 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: COPD; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: Participants will receive two different interventions after exertion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Vitabreath Device (Experimental): The Philips Respironics investigational device VitaBreath is a handheld, battery powered, intermittent positive airway pressure device that is non-invasive, and provides positive airway pressure (PAP) of 18 cm water (H2O) during inspiration and 8 cm H2O on expiration, thus creating 10 cm H2O of pressure support. Pressure support is defined as the difference between inhalation pressure and exhalation pressure. The study device is intended as an adjunct therapy to relieve shortness of breath in COPD patients who experience exertion-related dyspnea to allow them to be more active. The air is delivered to the patient via a mouthpiece on the device.
  Interventions: Device: Vitabreath Device
- Pursed Lip Breathing (Active Comparator): Pursed lip breathing is a commonly used technique by COPD patients. That involves exhaling through tightly pressed lips and inhaling through the nose with the mouth closed.
  Interventions: Other: Pursed Lip Breathing

INTERVENTIONS:
Device: Vitabreath Device — The VitaBreath device is designed for non-continuous use only and typical device use is expected to be for 2-3 minutes. The device should only be operated for less than 10 minutes at a time. After such time, the device should be turned off for at least 30 minutes
  Arms: Vitabreath Device
Other: Pursed Lip Breathing — Pursed lip breathing (PLB) is the standard of care and will be used as the control condition comparator.
  Arms: Pursed Lip Breathing

SUMMARY:
Dyspnea is the most common symptom limiting the ability of COPD patients to perform activities of daily living. Although there has been research involving the benefit of providing Non Invasive Ventilation (NIV) during exercise to increase tolerance overall, there is little research specifically looking at shortening dyspnea recovery times associated with exercise. We hypothesize that providing intermittent non-invasive positive pressure therapy (a form of NIV or PAP) with a handheld device to COPD patients immediately after exertion can relieve their dyspnea, and consequently allow them to be more active. In this study, we are comparing the distance walked as measured by a modified 6-Minute Walk Test (6MWT) of 20 COPD patients using VitaBreath (NIV) device versus Pursed Lip Breathing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40
* Ability to provide consent
* COPD diagnosis
* Forced Expiratory Volume in one second (FEV1) <55 and ≥ 25 percent of predicted value
* Perceived Shortness of Breath via the Modified Medical Research Counsel Dyspnea questionnaire (rating of 2 or greater) (Appendix B)
* Able to follow directions
* Able to tolerate mild physical activity
* Pursed Lip Breathing as standard of care
* No evidence of bullous lung disease (with any bullae greater than 3cm in diameter) as confirmed by a CT scan within the past one year.

Exclusion Criteria:

* Subjects who are acutely ill, medically complicated or who are medically unstable as determined by the investigator.
* Suffering from COPD exacerbation at time of enrollment or 60 days prior
* Subjects who are not currently prescribed oxygen and manifest oxygen desaturation below 88% on the screening 6MWT
* Subjects with heart disease or neuromuscular disease.
* Subjects who are not prescribed short-acting bronchodilator medication
* Patients who have experienced recent barotrauma or pneumothorax
* Unstable angina or Myocardial Infarction during past month
* Uncontrolled Hypertension (systolic blood pressure of >180mmHg (millimeters of Mercury) and a diastolic >100mmHg)
* Heart Rate >120 at rest
* Subjects who have trouble coordinating their breathing with the device during the device training, or cannot tolerate the device mouthpiece resulting in leaks from the nasal cavity
* Women of child-bearing potential (WOCP) who are pregnant, breast-feeding, or planning pregnancy during the course of the study. (WOCP must have a negative pregnancy test at every visit)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pullmonary Rehabilition Associates, Youngstown, Ohio
  - Pittsburgh Pulmonary Associates, Jefferson Hills, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Screened: All participants that were consented.
- Vitabreath First, Pursed Lip Breathing Second: The Philips Respironics investigational device VitaBreath is a handheld, battery powered, intermittent positive airway pressure device that is non-invasive, and provides positive airway pressure (PAP) of 18 cm water (H2O) during inspiration and 8 cm H2O on expiration, thus creating 10 cm H2O of pressure support. Pressure support is defined as the difference between inhalation pressure and exhalation pressure. The study device is intended as an adjunct therapy to relieve shortness of breath in COPD patients who experience exertion-related dyspnea to allow them to be more active. The air is delivered to the patient via a mouthpiece on the device.
- Pursed Lip Breathing First, Vitabreath Second: Pursed lip breathing is a commonly used technique by COPD patients. That involves exhaling through tightly pressed lips and inhaling through the nose with the mouth closed.
  Pursed Lip Breathing: Pursed lip breathing (PLB) is the standard of care and will be used as the control condition comparator.
Period: Screening
Arm/Group | Participants Screened | Vitabreath First, Pursed Lip Breathing Second | Pursed Lip Breathing First, Vitabreath Second
Started | 25 | 0 | 0
Completed | 20 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Screen Fail | 4 | 0 | 0
Not completed — Withdrawn | 1 | 0 | 0
Period: Intervention
Arm/Group | Participants Screened | Vitabreath First, Pursed Lip Breathing Second | Pursed Lip Breathing First, Vitabreath Second
Started | 0 | 10 | 10
Completed | 0 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants that were consented.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Body Mass Index (BMi) [Mean (Standard Deviation); unit: kg/m^2] — Population: One participant screen failed due to the results of their CT scan, and is therefore missing the baseline data that would have been collected after the scan.
  kg/m^2
    number analyzed (Participants) | 24
    (all) | 27.4 (6.7)
Heart Rate (bpm) [Mean (Standard Deviation); unit: beats per minute] — Population: One participant screen failed due to the results of their CT scan, and is therefore missing the baseline data that would have been collected after the scan
  beats per minute
    number analyzed (Participants) | 24
    (all) | 81.7 (16.6)
Systolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] — Population: One participant screen failed due to the results of their CT scan, and is therefore missing the baseline data that would have been collected after the scan
  mmHg
    number analyzed (Participants) | 24
    (all) | 136.1 (16.5)
Diastolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] — Population: One participant screen failed due to the results of their CT scan, and is therefore missing the baseline data that would have been collected after the scan
  mmHg
    number analyzed (Participants) | 24
    (all) | 78.5 (8.8)
FEV1(L) [Mean (Standard Deviation); unit: Liters] — Population: One participant screen failed due to the results of their CT scan, and is therefore missing the baseline data that would have been collected after the scan.
  Liters
    number analyzed (Participants) | 24
    (all) | 1.3 (0.6)
FEV1 (% Predicted) [Mean (Standard Deviation); unit: percentage of predicted FEV1] — Population: One participant screen failed due to the results of their CT scan, and is therefore missing the baseline data that would have been collected after the scan.
  percentage of predicted FEV1
    number analyzed (Participants) | 24
    (all) | 40.0 (16.8)
FVC (L) [Mean (Standard Deviation); unit: Liters] — Population: One participant screen failed due to the results of their CT scan, and is therefore missing the baseline data that would have been collected after the scan.
  Liters
    number analyzed (Participants) | 24
    (all) | 6.7 (22.0)
FVC (% Predicted) [Mean (Standard Deviation); unit: percentage of predicted FVC] — Population: One participant screen failed due to the results of their CT scan, and is therefore missing the baseline data that would have been collected after the scan.
  percentage of predicted FVC
    number analyzed (Participants) | 24
    (all) | 56.9 (13.2)
Pack Years [Mean (Standard Deviation); unit: packs per year] | 58.8 (31.4)

OUTCOME MEASURES:

1. Primary Outcome: Average Distance During Modified 6 Minute Walk Test
Description: Compare the average distance walked during modified 6 minute walk test (M 6MWT) by COPD participants using Pursed Lip Breathing (PLB) versus an intermittent positive airway pressure handheld device, VitaBreath.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Vitabreath Device | Pursed Lip Breathing
Number analyzed (Participants) | 20 | 20
meters
  1st Hallf of M 6MWT Distance | 128.0 (47.5) | 129.9 (43.3)
  2nd half of M 6MWT Distance | 137.5 (49.7) | 121.3 (38.9)
  Total M 6 MWT Distance | 265.5 (96.3) | 251.2 (80.8)
Statistical Analysis 1: Comparison: Vitabreath Device vs Pursed Lip Breathing; Test type: Superiority; p = 0.02, Wilcoxon Signed Rank — This p-value is in reference to the total Modified 6MWT Distance

ADVERSE EVENTS:
Time Frame: 1 Day
Groups:
- Vitabreath First, Pursed Lip Breathing Second: VitaBreath is a handheld, battery powered, intermittent positive airway pressure device that is non-invasive, and provides positive airway pressure (PAP) of 18 cm water (H2O) during inspiration and 8 cm H2O on expiration, thus creating 10 cm H2O of pressure support will be utilized first, followed by standard of care Pursed Lip Breathing.
- Pursed Lip Breathing First, Vitabreath Second: Pursed lip breathing (PLB) is the standard of care and will be used as the control condition comparator first followed by use of Vitabreath
Arm/Group | Participants Screened | Vitabreath First, Pursed Lip Breathing Second | Pursed Lip Breathing First, Vitabreath Second
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/25 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT03349437/Prot_SAP_000.pdf